CLINICAL TRIAL: NCT02013778
Title: Phase I-II Clinical Trial of the Safety and Preliminary Efficacy of Hydroxychloroquine Combined With Transarterial Chemoembolization in Unresectable Hepatocellular Carcinoma
Brief Title: Phase 1-2 Trial HCQ Plus TACE in Unresectable HCC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 22213
Record Dates: First submitted 2013-12-12; First posted 2013-12-17 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: outside of transplant criteria
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TACE + HCQ (Experimental): Subjects will receive HCQ plus standard of care TACE.
  Interventions: Drug: HCQ

INTERVENTIONS:
Drug: HCQ

SUMMARY:
Primary Phase I:To determine dose limiting toxicities and maximum tolerated dose (MTD) of the oral administration of hydroxychloroquine (HCQ) in conjunction with transarterial chemoembolization (TACE) in treating hepatocellular carcinoma (HCC). A conventional 3+3 design will be utilized. Primary Phase II: To evaluate the complete response rate in a cohort of patients treated at the MTD, A Simon's Optimal Two-stage design will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of giving informed consent
* Patient diagnosed with hepatocellular carcinoma in both lobes of the liver by one of the following methods (Pathologically confirmed HCC by biopsy or HCC 2 cm with classic radiographic findings of arterial phase enhancement with venous phase washout and pseudocapsule formation on contrast enhanced MRI or CT or Lesion greater than 2 cm with probable imaging features of HCC and imaging findings of cirrhosis and/or portal hypertension or a serum alphafetoprotein (AFP) greater than 200 mg/mL.
* Patient not candidate for orthotopic liver transplantation at the Hospital of the University of Pennsylvania based on review of patient imaging and history at multidisciplinary Hepatic Tumor Conference at the Hospital of the University of Pennsylvania.
* Age 18 years old
* Albumin 2.4 g/dL; Total bilirubin 2 mg/dL; INR 1.5
* Creatinine 2.0 mg/dL, AST 121 IU/L; ALT 189 IU/L
* Child-Turcotte-Pugh Classification A or B
* Eastern Clinical Oncology Group performance status 0 or1.

Exclusion Criteria:

* Prior TACE
* Active GI hemorrhage within 2 weeks of study enrollment
* Ascites refractory to medical therapy
* Contraindication to receiving HCQ or TACE
* Unilobar HCC
* Contraindication to contrast enhanced MRI (i.e. unable to undergo follow-up imaging)
* Women who are pregnant
* Participation in another concurrent treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Nadolski, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TACE + HCQ: Subjects will receive Hydroxychloroquine (HCQ) plus standard of care Transarterial Chemoembolization (TACE).
Period: Overall Study
Arm/Group | TACE + HCQ
Started | 8
Completed | 1
Not Completed | 7
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- TACE + HCQ: Subjects will receive HCQ plus standard of care TACE.
  HCQ
Arm/Group | TACE + HCQ
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Bilobar Hepatocellular Cancer (HCC) [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse Events graded according to the Common Terminology Criteria of Adverse Events (CTCAE) version 4.0
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TACE + HCQ
Number analyzed (Participants) | 8
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 year
Description: All adverse events occurring during the study period (up to 6 months after last dose of HCQ) were recorded. The clinical course of each event was followed until resolution, stabilization, or until it was determined that the study treatment or participation is not the cause. Serious adverse events that were still ongoing at the end of the study period must be followed up to determine the final outcome.
Arm/Group | TACE + HCQ
All-Cause Mortality (participants affected / at risk) | 7/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TACE + HCQ (N=8)
Pain (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT02013778/Prot_SAP_ICF_000.pdf